CLINICAL TRIAL: NCT02807714
Title: Role of Podocan and Wnt Pathway Regulatory Molecules in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Jennifer Victory, RN, CCRC (Other)
Collaborators: Baylor University (Other)
Responsible Party: Sponsor-Investigator, Jennifer Victory, RN, CCRC, Clinical Research Nurse Supervisor, Bassett Healthcare
Organization: Bassett Healthcare (Other)
Other Study IDs: 2042
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- No CAD: Patients scheduled for elective cardiac catheterization for evaluation of suspected CAD that are found to not have CAD
- Obstructive CAD (non-ACS) Group: Patients scheduled for elective cardiac catheterization for evaluation of known or suspected CAD that are found to have obstructive CAD requiring intervention.
- Stable CAD, no intervention required: Patients scheduled for elective cardiac catheterization for evaluation of known or suspected CAD that are found to have non-obstructive CAD not requiring intervention.
- Acute Coronary Syndrome (ACS): Patients who undergo an emergent cardiac catheterization for evaluation of known or suspected STEMI, NSTEMI, Unstable Angina (UA).

SUMMARY:
The purpose of this study is to find an association between a protein named Podocan and WNT pathway regulatory molecules in patients with different forms of Coronary Artery Disease (Acute Coronary syndrome, Stable Angina and Coronary Artery Restenosis). It has been found in experimental studies that this protein is regulating smooth muscle cell function and hence may be influencing the progression of Coronary Artery Disease (CAD). We are testing to see if the same regulatory function exists in human subjects. Studying patient's blood will possibly enable to identify an association between Podocan and CAD. This may help to better prevent and treat CAD with improved understanding of the mechanism of the disease. No drugs or other therapeutic interventions will be used for the purpose of the research study. Only blood samples will be collected in the cardiac catheterization lab. As a part of this study participants will be followed for repeat events or repeat cardiac catheterization over a period of 24 months.

DETAILED DESCRIPTION:
Smooth muscle cells (SMC's) critically influence the clinical course of vascular disease . The close regulation of SMC migration and proliferation within the intimal space is critical in maintaining a delicate balance between insufficient and excessive atherosclerotic plaque repair . When SMC proliferation is too suppressed, the ensuing weakening of the fibrous cap can result in plaque vulnerability underlying Acute Coronary Syndrome and when SMC proliferation is excessive, intimal hyperplasia as hallmark of accelerated Coronary Artery Disease can follow such as in Restenosis post PCI. While stents have vastly improved upon the recoil and constrictive remodeling component of restenosis, the problem of accelerated intimal SMC growth has remained. The current approach of delivering stents releasing non-specific agents promoting cell death and/or inhibition of proliferation has been successful at lowering the need for recurrent vascular interventions . However, this success comes at the expense of delaying vascular healing, whose ultimate long-term clinical impact is still being evaluated. Short and long-term negative effects on the healing arterial wall such as delayed re-endothelialization, increased inflammation and enhanced thrombogenicity of drug-eluting stent (DES) are undisputed. These side effects of DES are being masked by prolonged and aggressive dual anti-platelet therapy, which is exposing patients - especially the elderly - to increased bleeding risks and complicates clinical decision-making. This problem also causes fear of too early treatment cessation, demands rigorous patient compliance and is costly. These issues are not trivial in daily clinical practice and the lack of reliable clinical predictors of restenosis precludes individualized and patient tailored stent selection.

Podocan is a protein within the Single Leucine Rich (SLR) protein family and is a previously unrecognized component of the sclerotic glomerular lesion that develops in the course of experimental HIV associated nephropathy . Its important role in regulating smooth muscle cell function via the Wnt-pathway has been recently described by the investigators of this study . It has been shown to modulate experimental arterial repair and a significantly different expression pattern has been found in coronary arterial lesions obtained by directional coronary atherectomy (DCA) from patients with restenosis compared to stable angina . These findings do suggest a possible clinical predictive role of Podocan, and the Wnt-pathway effectory molecules on the incidence of Instent Re-stenosis (ISR) and the need for Repeat Target Vessel Revascularization.

All patients who present to the cardiac cath lab for angiography for the evaluation of known or suspected CAD will be eligible for enrollment. It is expected that, based on angiographic results, participants will fall into one of four categories:

1. No CAD
2. Stable CAD, no intervention required
3. Obstructive CAD requiring intervention (angioplasty, stenting, CABG) (Not associated with acute event, such as MI)
4. Patients presenting with Acute Coronary Syndrome (ACS)

   In all elective/scheduled case, prior to catheterization, a peripheral blood sample will be obtained via an IV access line previously placed for the catheterization procedure. In emergent cases of ACS, blood samples will be obtained in the same manner described previously if possible. It is likely that in some cases, such as ST elevation myocardial infarction (STEMI), this will not be possible based on clinical care priorities. In these cases blood samples will be obtained within 24 hours after catheterization. These blood samples will need to be obtained via venipuncture and will be clearly labeled/recorded as being collected post-procedure. Blood samples will be frozen and stored in a -80°C freezer in the Research Institute. Samples will be batch sent to Baylor Medical Center to be tested for the presence of Wnt and Podocan molecules (Wnt-1, Wnt-3, Dkk-1, Sclerostin, WIF-1, sFRP-1, sFRP-3) by measuring circulating levels via ELISA Obstructive CAD (non-ACS) Group: It is expected that 900 stented patients will be enrolled over 18-20 months. Justification of patient numbers is derived by specific aim of attempting to establish prospective component of our study, which is the prediction of restenosis. Given a current average incidence of restenosis between 10 to 15 % (DES around 7% and BMS around 20% restenosis rate) this number should guarantee around 100 restenosis events out of 900 patients. This should give a realistic statistical chance to detect a possible clinical predictive value of our variables. Participants who are consented and sampled but who are found not to have obstructive CAD requiring stenting will be maintained separately in the study database as a control group for future analysis.

   The following information will be collected from the baseline angiogram:
   * syntax score in order to determine the coronary atherosclerotic burden
   * PCI performed during baseline angiogram? If yes - what type of stent, location

   Participant charts will be reviewed at 24 months post catheterization to collect covariates (like age, sex, race/ethnicity, high blood pressure, obesity, smoking and diabetes) and to monitor for the following events:
   * Repeat cardiac catheterization

     --Re-stenosis of stent placed at baseline angiogram

     --Onset of new lesions
     * Progression of lesions not treated at baseline angiogram
   * New onset MI/ACS
   * Recurrent MI/ACS
   * Death due to known cardiovascular causation

   CS Group:

   The following information will be collected from the baseline angiogram:
   * syntax score in order to determine the coronary atherosclerotic burden
   * PCI performed during baseline angiogram? If yes - what type of stent, location

   Participant charts will be reviewed at 24 months post catheterization to monitor for the following events:
   * Repeat cardiac catheterization --Re-stenosis of stent placed at baseline angiogram

     --Onset of new lesions

     --Progression of lesions not treated at baseline angiogram
   * Recurrent MI/ACS
   * Death due to known cardiovascular causation

   Non- Obstructive/Stable CAD Group:

   The following information will be collected from the baseline angiogram:

   -syntax score in order to determine the coronary atherosclerotic burden

   Participant charts will be reviewed at 24 months post catheterization to monitor for the following events:
   * Repeat cardiac catheterization

     --Onset of new lesions

     --Progression of lesions not treated at baseline angiogram
   * New onset MI/ACS
   * Death due to known cardiovascular causation

   Normal Angiography (No CAD) Group:

   Participant charts will be reviewed at 24 months post catheterization to monitor for the following events:
   * Repeat cardiac catheterization --Onset of new lesions

     * Progression of lesions not treated at baseline angiogram
   * New onset MI/ACS
   * Death due to known cardiovascular causation

   Comparison with Historical Samples: The principal investigator owns a collection of historical tissue samples that have angiographically defined coronary target lesion biopsies from clinical patients with stable angina and restenosis. The technique of DCA (Directional Coronary Artherectomy), by which these samples were collected, is not clinically done anymore, preventing the investigators from collecting these samples from the current study participants. The current study participants will be grouped according to exact same clinical criteria as the historic patients and hence represent comparable clinical cohort. The expression of Podocan and Wnt effectory molecules (Wnt-1, Wnt-3, Dkk-1, Sclerostin, WIF-1, sFRP-1, sFRP-3) in coronary artery lesions obtained by Directional Coronary Artherectomy will be analyzed using immuno-histochemical staining and quantitative histo-morphometric analysis comparing restenosis with Primary Stable Coronary Artery Disease as published by the investigators (5). This comparison will allow the investigators to examine the relationship between the level of the Podocan and Wnt effectory molecules, coronary plaque physiology, and the study endpoint of disease progression as evidenced by restenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Scheduled for coronary angiography in the cardiac catheterization lab
* Able to provide informed consent

Exclusion Criteria:

* Previously enrolled & sampled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective cardiac catheterization for known or suspected CAD.
Sampling Method: Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Podocan levels | Day 1
  Prior to catheterization, a peripheral blood sample will be obtained via an IV access line previously placed for the catheterization procedure. Blood samples will be frozen and stored in a -80°C freezer in the Research Institute.
WNT regulatory molecules | Day1
  Prior to catheterization, a peripheral blood sample will be obtained via an IV access line previously placed for the catheterization procedure. Blood samples will be frozen and stored in a -80°C freezer in the Research Institute.

SECONDARY OUTCOMES:
Restenosis | 24 months
Onset of new lesions | 24 months
progression of existing lesions | 24 months
New onset MI/ACS | 24 months
Death due to known cardiovascular causation | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Randolph Hutter, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided